CLINICAL TRIAL: NCT00124176
Title: Continuous Levalbuterol for Treatment of Status Asthmaticus in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #2004-12-4130
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2012-12

CONDITIONS: Asthma
Keywords: Asthma; Levalbuterol; Albuterol; Children
MeSH Terms: conditions — Asthma | interventions — Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Nebulized levalbuterol 10mg/hr given continuously
  Interventions: Drug: Levalbuterol (R albuterol)
- 2 (Active Comparator): Racemic albuterol 20mg/hr given continuously
  Interventions: Drug: Racemic albuterol (R+S albuterol)

INTERVENTIONS:
Drug: Racemic albuterol (R+S albuterol) — 20mg/hr continuous racemic albuterol
  Arms: 2
Drug: Levalbuterol (R albuterol) — 10mg/hr continuous nebulized levalbuterol
  Other Names: Xopenex
  Arms: 1

SUMMARY:
This study will use a randomized, double-blind, controlled trial design in order to assess the safety and efficacy of levalbuterol (LEV) compared to racemic albuterol (RAC) when delivered continuously in a high-dose regimen for children with severe exacerbations of asthma.

Primary hypothesis

* Children with severe asthma receiving continuous levalbuterol will have a shorter duration of continuous therapy as compared to racemic albuterol.

Secondary hypotheses

* Children receiving continuous levalbuterol will have improved lung function measured by forced expiratory volume at 1 second (FEV1) as compared to racemic albuterol.
* Children receiving continuous levalbuterol will have improved clinical asthma score as compared to racemic albuterol.

DETAILED DESCRIPTION:
High-dose nebulized albuterol is standard therapy for severe asthma exacerbations at The Children's Hospital of Philadelphia (CHOP) and other tertiary care pediatric hospitals throughout the United States. For the most severe exacerbations, albuterol is provided continuously at high doses until improvement is observed. This regimen has been standardized in a treatment protocol that has been used at CHOP for more than 5 years. Recently, levalbuterol (LEV), the purified active (R)-enantiomer of albuterol, has been approved for use in acute asthma. Preliminary evidence suggests that LEV may improve pulmonary function and clinical outcomes in children with asthma based on studies using standard dosing regimens. Laboratory and clinical evidence suggest that the (S)-enantiomer of albuterol may have detrimental effects that contribute to poor response to racemic albuterol (RAC). Limited data exist about the efficacy of LEV in high-dose regimens.

This study will use a randomized, double-blind, controlled trial design in order to assess the safety and efficacy of LEV compared to RAC when delivered continuously in a high-dose regimen for severe exacerbations of asthma. Children treated for asthma exacerbations in the CHOP emergency department (ED) will be eligible for study enrollment. Those that meet enrollment criteria will be randomized to receive either high dose RAC according to the standard asthma care protocol or equivalent dosing of LEV. Approximately 128 patients with 64 in each arm of the study will be enrolled. An interim safety analysis will be conducted after the first 40 patients are enrolled. This study should be completed in six to nine months. The primary outcome will be duration of continuous therapy. Secondary outcomes will include improvement of clinical asthma score and change in forced expiratory volume in one second (FEV1). In addition, (R)-albuterol and (S)-albuterol levels will be measured at study entry and at 6-hour intervals in the first 40 patients enrolled. These values will be used to determine prior RAC exposure and to determine serum levels of (R) and (S) albuterol during continuous therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years of age
* Diagnosis of asthma with two previous visits to emergency department (ED) or primary care provider for asthma care
* Clinical decision by ED attending physician to begin continuous albuterol after standardized initial ED treatment.

Exclusion Criteria:

* Clinical decision to begin continuous intravenous beta-agonist infusion (e.g. terbutaline)
* Clinical decision to admit to the Pediatric Intensive Care Unit
* Drug allergy or other contraindication to RAC or LEV
* Other concurrent disease such as sickle cell disease, cystic fibrosis, or cardiac disease
* Pregnancy
* Prior enrollment in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2004-04; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Zorc, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Levalbuterol (R) Nebulized Solution: Continuous levalbuterol nebulized solution 10mg/hr given as continuous nebulization
- Continuous Racemic (R+S) Albuterol: Continuous racemic albuterol 20mg/hr given as continuous nebulization
Period: Overall Study
Arm/Group | Continuous Levalbuterol (R) Nebulized Solution | Continuous Racemic (R+S) Albuterol
Started | 40 | 41
Received Study Drug | 37 (3 never started on drug due to improvement but were kept in the study by intention to treat.) | 41
Completed | 40 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Levalbuterol (R) Nebulized Solution | Continuous Racemic (R+S) Albuterol | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 41 | 81
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.4 (3.5) | 10.7 (3.3) | 10.6 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 26 | 25 | 51
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Duration of Continuous Therapy
Description: standard intention to treat (ITT) analysis
Time Frame: During hospitalization
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Continuous Levalbuterol (R) Nebulized Solution | Continuous Racemic (R+S) Albuterol
Number analyzed (Participants) | 40 | 41
Hours | 18.3 [11 to 25] | 16 [11 to 25]

2. Secondary Outcome: Change in Pediatric Asthma Severity Score
Description: Change in Pediatric Asthma Severity Score. Range 0 (best) - 6 (worst)
  Score at each time point is calculated by adding 3 elements:
  Wheeze (0= None/Mild, 1=Moderate, 2=Severe) Prolonged expiration (0= None/Mild, 1=Moderate, 2=Severe) Work of breathing (0= None/Mild, 1=Moderate, 2=Severe)
Time Frame: After 12 hours of continuous nebulization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Levalbuterol (R) Nebulized Solution | Continuous Racemic (R+S) Albuterol
Number analyzed (Participants) | 40 | 41
units on a scale | -1.0 (1.2) | -0.64 (1.7)

3. Secondary Outcome: Heart Rate
Time Frame: After 12 hours of continuous nebulization
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Continuous Levalbuterol (R) Nebulized Solution | Continuous Racemic (R+S) Albuterol
Number analyzed (Participants) | 40 | 41
beats per minute | 132 (16.4) | 132 (18.4)

4. Secondary Outcome: Serum Potassium Levels
Time Frame: After 12 hours of continuous nebulization
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Continuous Levalbuterol (R) Nebulized Solution | Continuous Racemic (R+S) Albuterol
Number analyzed (Participants) | 40 | 41
mg/dL | 3.6 (0.6) | 3.6 (0.4)

5. Secondary Outcome: Serum Albuterol S Isomer Levels
Time Frame: After 6 hours of continuous albuterol
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Continuous Levalbuterol (R) Nebulized Solution | Continuous Racemic (R+S) Albuterol
Number analyzed (Participants) | 40 | 41
ng/mL | 5.5 (3.3) | 28.6 (11.7)

ADVERSE EVENTS:
Arm/Group | Continuous Levalbuterol (R) Nebulized Solution | Continuous Racemic (R+S) Albuterol
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No